CLINICAL TRIAL: NCT03863015
Title: Interleukin-6 Receptor Antibodies for Modulating the Systemic Inflammatory Response After Out-of-Hospital Cardiac Arrest - a Randomized Clinical Trial
Brief Title: IL-6 Inhibition for Modulating Inflammation After Cardiac Arrest
Acronym: IMICA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Hassager (Other)
Responsible Party: Sponsor-Investigator, Christian Hassager, Professor, MD, DMSc, FESC, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT:2018-002686-19
Record Dates: First submitted 2019-02-22; First posted 2019-03-05 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Heart Arrest; Out-Of-Hospital Cardiac Arrest; Systemic Inflammatory Response Syndrome
Keywords: OHCA; PCAS; SIRS; Inflammation; RoActemra; Tociluzumab
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest; Systemic Inflammatory Response Syndrome; Inflammation | interventions — tocilizumab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 fashion to receive IL-6RA or placebo. Patients being allocated to IL-6RA will receive a one-hour infusion of 8 mg tocilizumab per kg body weight (maximum dose 800 mg, 40 mL), equivalent to 0.4 mL per kg bodyweight (study drug concentration 20 mg/mL). Patients being allocated to placebo will receive a one-hour infusion of 0.4 mL /kg body weight of normal saline (maximum dose 40 mL)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Active Comparator): A one hour infusion of a single 8mg/kg dose (max. 800mg) of tocilizumab to attenuate systemic inflammation after out-of-hospital cardiac arrest, given as early as possible after hospital admission.
  Interventions: Drug: Tocilizumab 20 Mg/mL Intravenous Solution
- Isotonic saline (Placebo Comparator): A one hour infusion of isotonic saline
  Interventions: Drug: isotonic saline

INTERVENTIONS:
Drug: Tocilizumab 20 Mg/mL Intravenous Solution — Tocilizumab is suspended in isotonic saline to a total volume of 100mL prior to infusion
  Other Names: RoActemra
  Arms: Tocilizumab
Drug: isotonic saline — A one hour infusion of 100mL isotonic saline
  Other Names: Placebo
  Arms: Isotonic saline

SUMMARY:
Resuscitated cardiac arrest is associated with a systemic inflammatory response that is directly associated with poor prognosis. Inhibition of the IL-6 mediated immune response may potentially inhibit the systemic inflammatory response, potentially improving the prognosis of these severely ill patients.

DETAILED DESCRIPTION:
INTRODUCTION AND BACKGROUND:

The incidence of out-of-hospital cardiac arrest (OHCA) in Denmark is approximately 4,000 per year, and the mortality remains approximately 90%. Furthermore, in the approximately 30% of patients who are resuscitated and admitted to the intensive care unit (ICU), the mortality within the first month remains between 50% to 70%. Accordingly, an increasing emphasis on post-resuscitation care has been addressed by contemporary guidelines.

The high mortality after resuscitated OHCA has been attributed to a post-cardiac arrest syndrome (PCAS), which includes four mutually interacting components: a systemic inflammatory response (SIRS)-like syndrome, cerebral injury, myocardial dysfunction, and the persistent precipitating cause of the arrest. Despite repeated emphasis on post-resuscitation care, no specific therapies targeting PCAS have been implemented, with the exception of targeted temperature management (TTM), which has been recommended since 2003. Accordingly, research addressing mitigation of the PCAS seems intuitively beneficial.

During and after OHCA, exposure to whole-body ischemia and reperfusion injury triggers activation of inflammatory cascades leading to a sepsis-like syndrome. A multitude of inflammatory markers have been associated with unfavorable outcome after OHCA, including procalcitonin (PCT), c-reactive protein (CRP), interleukin (IL) 6, and IL-10.

Furthermore, the inflammatory markers interleukin 1β (IL-1β), IL-6, IL-10, and tumor necrosis factor α (TNF-α) have all been associated with the severity of PCAS, assessed by sequential organ failure assessment (SOFA) score. Importantly, levels of IL-6 have been shown to be independently associated with unfavorable outcome after adjustment for known risk markers. Further, the level of IL-6 was more strongly associated with PCAS severity compared to classical inflammatory markers such as CRP and PCT.

Interleukin-6 is a pro-inflammatory cytokine secreted by T cells and macrophages. IL-6 readily crosses the blood-brain-barrier and is a mediator of fever. Further, IL-6 is a mediator of the acute phase response and plays a role in activation of the coagulation system, increasing vascular permeability, and weakening papillary muscle contractions leading to myocardial dysfunction. As such, IL-6 is involved in pathological processes including tissue hypoxia, disseminated intravascular coagulation (DIC), and multiorgan failure, all of which represent parts of the SIRS response. IL-6 has been suggested to play a role in ischemia-reperfusion injury in myocardial infarction (MI), and higher levels of IL-6 have been associated both with the magnitude of myocardial injury, mortality and adverse events in this group.

Due to the role of IL-6 in many inflammatory diseases, IL-6 receptor antibodies (IL-6RA) have been developed. The first IL-6RA, tocilizumab, was approved for treatment of rheumatoid arthritis in 2009, and has later been approved for giant cell arthritis and chimeric antigen receptor (CAR) T cell-induced cytokine release syndrome. In addition to the approved indications, tocilizumab has been suggested to have other beneficial immune modulating and organ protective effects.

In patients presenting with non-ST-elevation myocardial infarction (NSTEMI), a one-hour infusion of 280mg tocilizumab decreased the inflammatory response assessed by CRP levels, and further decreased myocardial injury assessed by TnT levels. Importantly, no increased risk of adverse events was observed in patients receiving tocilizumab. Animal data suggest that tocilizumab is safe and effective for treatment of severe acute pancreatitis and associated acute lung injury. Further, tocilizumab had neuroprotective effects in a model of Alzheimer disease. In humans, tocilizumab has been suggested to be effective against the autoimmune neurological disorders neuromyelitis optica and autoimmune encephalitis.

In summary, resuscitated OHCA is associated with a severe SIRS-like response, the magnitude of which has been associated with increased mortality and poor neurological outcome. Inhibiting the IL-6 mediated immune response may inhibit the SIRS-like response and may further inhibit ischemia-reperfusion injury leading to improved outcome.

HYPOTHESIS:

A one-hour infusion of the IL-6RA tocilizumab initiated as soon as possible after ROSC will reduce the SIRS-like response assessed by hsCRP levels after OHCA.

SAMPLE SIZE:

A total of 80 patients will be included, i.e. 40 being allocated to IL-6RA and placebo, respectively. Patients who die or become hemodynamically unstable immediately after randomization before the study drug has been prepared will be excluded from the modified intention to treat population and replaced by randomizing additional patients. Likewise, patients for whom the relatives refuse study participation when informed of the study and asked for consent (before the patients can be asked) will be excluded from the modified intention to treat population and replaced.

ELIGIBILITY:
Inclusion Criteria:

Each of the following criteria must be fulfilled for a subject to be eligible:

1. Age ≥ 18 years
2. OHCA of a presumed cardiac cause
3. Unconsciousness upon admission, i.e. a GCS < 9
4. Sustained ROSC for more than 20 minutes

Exclusion Criteria:

None of the following criteria must be fulfilled for a subject to be eligible:

1. Consciousness upon admission, i.e. a GCS ≥ 9
2. Presumed non-cardiac cause of arrest
3. Unwitnessed asystole
4. Suspected or confirmed intracranial bleeding or stroke
5. Pregnancy, or females in fertile age, unless a negative serum HCG can rule out pregnancy within the inclusion window.
6. Temperature on admission < 30 °C
7. Persistent cardiogenic shock* that is not reversed within the inclusion window
8. Known disease making 180 day survival unlikely
9. Known limitations in therapy
10. Known pre-arrest Cerebral Performance Category of 3 to 4
11. > 240 minutes from ROSC to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Concentration of hsCRP | Daily measurements from admission to 72 hours after admission.
  high sensitivity C-reactive protein

SECONDARY OUTCOMES:
Biomarkers of organ damage | Plasma/serum samples and routine biochemistry are collected at admission, 24h, 48h and 72h (NSE only at 48 and 72h)
  Markers of cerebral injury: Neuron-specific enolase (NSE) levels (routine biochemistry), and other markers of cerebral injury (analysis of samples in biobank).
  Markers of cardiac injury: Troponin T (TnT) and CKMB levels. Markers of kidney injury: Creatinine levels. Markers of hepatic injury: ALAT, ASAT, bilirubin, INR. Markers of endothelial injury: soluble thrombomodulin levels.
Markers of inflammation, interleukin levels | At admission, 24h, 48h & 72h
  Interleukin levels: INF-g, IL-1b, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8 IL-10, IL-12, IL-13, IL-17A, G-CSF, GM-CSF, MCP-1 og MIP-1beta and TNF-α (analysis of samples in biobank).
Markers of inflammation, leukocytes | At admission, 24h, 48h & 72h
  Leukocyte differential count.
Markers of inflammation, SOFA score | The first 3 days from admission
  Daily Sequential Organ Failure Assessment (SOFA) scores.
Markers of the coagulation system, fibrinogen | At admission, 48h and 72h
  The possible downstream effect of dampened inflammation on the coagulation system is evaluated by the concentration of plasma-fibrinogen.
Markers of the coagulation system, thrombelastography | At admission and 48h
  The possible downstream effect of dampened inflammation on the coagulation system is evaluated by whole blood thrombelastography.
Markers of hemodynamic function, Swan-Ganz Catheter | At admission, 24h, 48h & 72h
  Swan-Ganz based measurements of cardiac output, central venous pressure, pulmonary capillary wedge pressure, and systemic vascular resistance.
Markers of hemodynamic function, Arterial blood gasses | At admission, 2h, 4h, 6h, 8h, 10h, 12h, 18h, 24h, 30h, 36h, 48h, 72h, 96h and 120h (sampling ceases if the arterial line is discontinued).
  Arterial blood gasses including lactate and base excess at frequent intervals.
Markers of hemodynamic function, Echocardiography | Day 1 and on either day 3, 4 or 5.
  Transthoracic echocardiography including assesment of left ventricular ejection fraction (LVEF) and tricuspid annular plane systolic excursion (TAPSE).
Clinical endpoints, Survival | At 30 days, 90 days, 180 days, and at end of trial.
  Survival.
Clinical endpoints, MOCA score | At 90 days.
  Montreal Cognitive Assessment (MOCA) score at 90 days.
Clinical endpoints, CPC | At 30 days, 90 days and 180 days.
  Cerebral Performance Category (CPC) at 30 days, 90 days and 180 days, assessed by telephone interview and/or review of medical file after completion of the 180 days.
Safety: incidence of adverse events | From admission till 7 days.
  Cumulated incidence of adverse events the first 7 days.

OTHER OUTCOMES:
Predefined sub-study: MRI of heart and brain | The day following admission.
  A subset of the trial participants will be enrolled in a sub-study focusing on cardio protection and neuroprotection as a pilot investigation. This sub-study will include an echocardiography, a cerebral MR scan and a cardiac MR scan; all three modalities being performed the day following admission.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hassager, MD, DMSc, Principal Investigator — Department of Cardiology, The Heart Center, Rigshospitalet, Copenhagen, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wissenberg M, Lippert FK, Folke F, Weeke P, Hansen CM, Christensen EF, Jans H, Hansen PA, Lang-Jensen T, Olesen JB, Lindhardsen J, Fosbol EL, Nielsen SL, Gislason GH, Kober L, Torp-Pedersen C. Association of national initiatives to improve cardiac arrest management with rates of bystander intervention and patient survival after out-of-hospital cardiac arrest. JAMA. 2013 Oct 2;310(13):1377-84. doi: 10.1001/jama.2013.278483. PMID 24084923
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Soholm H, Wachtell K, Nielsen SL, Bro-Jeppesen J, Pedersen F, Wanscher M, Boesgaard S, Moller JE, Hassager C, Kjaergaard J. Tertiary centres have improved survival compared to other hospitals in the Copenhagen area after out-of-hospital cardiac arrest. Resuscitation. 2013 Feb;84(2):162-7. doi: 10.1016/j.resuscitation.2012.06.029. Epub 2012 Jul 13. PMID 22796541
- [Background] Callaway CW, Donnino MW, Fink EL, Geocadin RG, Golan E, Kern KB, Leary M, Meurer WJ, Peberdy MA, Thompson TM, Zimmerman JL. Part 8: Post-Cardiac Arrest Care: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S465-82. doi: 10.1161/CIR.0000000000000262. No abstract available. PMID 26472996
- [Background] Nolan JP, Soar J, Cariou A, Cronberg T, Moulaert VR, Deakin CD, Bottiger BW, Friberg H, Sunde K, Sandroni C. European Resuscitation Council and European Society of Intensive Care Medicine Guidelines for Post-resuscitation Care 2015: Section 5 of the European Resuscitation Council Guidelines for Resuscitation 2015. Resuscitation. 2015 Oct;95:202-22. doi: 10.1016/j.resuscitation.2015.07.018. No abstract available. PMID 26477702
- [Background] Neumar RW, Nolan JP, Adrie C, Aibiki M, Berg RA, Bottiger BW, Callaway C, Clark RS, Geocadin RG, Jauch EC, Kern KB, Laurent I, Longstreth WT Jr, Merchant RM, Morley P, Morrison LJ, Nadkarni V, Peberdy MA, Rivers EP, Rodriguez-Nunez A, Sellke FW, Spaulding C, Sunde K, Vanden Hoek T. Post-cardiac arrest syndrome: epidemiology, pathophysiology, treatment, and prognostication. A consensus statement from the International Liaison Committee on Resuscitation (American Heart Association, Australian and New Zealand Council on Resuscitation, European Resuscitation Council, Heart and Stroke Foundation of Canada, InterAmerican Heart Foundation, Resuscitation Council of Asia, and the Resuscitation Council of Southern Africa); the American Heart Association Emergency Cardiovascular Care Committee; the Council on Cardiovascular Surgery and Anesthesia; the Council on Cardiopulmonary, Perioperative, and Critical Care; the Council on Clinical Cardiology; and the Stroke Council. Circulation. 2008 Dec 2;118(23):2452-83. doi: 10.1161/CIRCULATIONAHA.108.190652. Epub 2008 Oct 23. No abstract available. PMID 18948368
- [Background] Nolan JP, Morley PT, Vanden Hoek TL, Hickey RW, Kloeck WG, Billi J, Bottiger BW, Morley PT, Nolan JP, Okada K, Reyes C, Shuster M, Steen PA, Weil MH, Wenzel V, Hickey RW, Carli P, Vanden Hoek TL, Atkins D; International Liaison Committee on Resuscitation. Therapeutic hypothermia after cardiac arrest: an advisory statement by the advanced life support task force of the International Liaison Committee on Resuscitation. Circulation. 2003 Jul 8;108(1):118-21. doi: 10.1161/01.CIR.0000079019.02601.90. No abstract available. PMID 12847056
- [Background] Adrie C, Laurent I, Monchi M, Cariou A, Dhainaou JF, Spaulding C. Postresuscitation disease after cardiac arrest: a sepsis-like syndrome? Curr Opin Crit Care. 2004 Jun;10(3):208-12. doi: 10.1097/01.ccx.0000126090.06275.fe. PMID 15166838
- [Background] Adrie C, Adib-Conquy M, Laurent I, Monchi M, Vinsonneau C, Fitting C, Fraisse F, Dinh-Xuan AT, Carli P, Spaulding C, Dhainaut JF, Cavaillon JM. Successful cardiopulmonary resuscitation after cardiac arrest as a "sepsis-like" syndrome. Circulation. 2002 Jul 30;106(5):562-8. doi: 10.1161/01.cir.0000023891.80661.ad. PMID 12147537
- [Background] Fries M, Kunz D, Gressner AM, Rossaint R, Kuhlen R. Procalcitonin serum levels after out-of-hospital cardiac arrest. Resuscitation. 2003 Oct;59(1):105-9. doi: 10.1016/s0300-9572(03)00164-3. PMID 14580740
- [Background] Stammet P, Devaux Y, Azuaje F, Werer C, Lorang C, Gilson G, Max M. Assessment of procalcitonin to predict outcome in hypothermia-treated patients after cardiac arrest. Crit Care Res Pract. 2011;2011:631062. doi: 10.1155/2011/631062. Epub 2011 Oct 26. PMID 22110909
- [Background] Bro-Jeppesen J, Kjaergaard J, Wanscher M, Nielsen N, Friberg H, Bjerre M, Hassager C. Systemic Inflammatory Response and Potential Prognostic Implications After Out-of-Hospital Cardiac Arrest: A Substudy of the Target Temperature Management Trial. Crit Care Med. 2015 Jun;43(6):1223-32. doi: 10.1097/CCM.0000000000000937. PMID 25756419
- [Background] Bro-Jeppesen J, Kjaergaard J, Wanscher M, Nielsen N, Friberg H, Bjerre M, Hassager C. The inflammatory response after out-of-hospital cardiac arrest is not modified by targeted temperature management at 33 degrees C or 36 degrees C. Resuscitation. 2014 Nov;85(11):1480-7. doi: 10.1016/j.resuscitation.2014.08.007. Epub 2014 Aug 19. PMID 25150183
- [Background] Banks WA, Kastin AJ, Gutierrez EG. Penetration of interleukin-6 across the murine blood-brain barrier. Neurosci Lett. 1994 Sep 26;179(1-2):53-6. doi: 10.1016/0304-3940(94)90933-4. PMID 7845624
- [Background] Tanaka T, Narazaki M, Kishimoto T. Interleukin (IL-6) Immunotherapy. Cold Spring Harb Perspect Biol. 2018 Aug 1;10(8):a028456. doi: 10.1101/cshperspect.a028456. PMID 28778870
- [Background] Sawa Y, Ichikawa H, Kagisaki K, Ohata T, Matsuda H. Interleukin-6 derived from hypoxic myocytes promotes neutrophil-mediated reperfusion injury in myocardium. J Thorac Cardiovasc Surg. 1998 Sep;116(3):511-7. doi: 10.1016/S0022-5223(98)70018-2. PMID 9731794
- [Background] Zamani P, Schwartz GG, Olsson AG, Rifai N, Bao W, Libby P, Ganz P, Kinlay S; Myocardial Ischemia Reduction with Aggressive Cholesterol Lowering (MIRACL) Study Investigators. Inflammatory biomarkers, death, and recurrent nonfatal coronary events after an acute coronary syndrome in the MIRACL study. J Am Heart Assoc. 2013 Jan 28;2(1):e003103. doi: 10.1161/JAHA.112.003103. PMID 23525424
- [Background] Lopez-Cuenca A, Manzano-Fernandez S, Lip GY, Casas T, Sanchez-Martinez M, Mateo-Martinez A, Perez-Berbel P, Martinez J, Hernandez-Romero D, Romero Aniorte AI, Valdes M, Marin F. Interleukin-6 and high-sensitivity C-reactive protein for the prediction of outcomes in non-ST-segment elevation acute coronary syndromes. Rev Esp Cardiol (Engl Ed). 2013 Mar;66(3):185-92. doi: 10.1016/j.rec.2012.07.019. Epub 2012 Dec 8. PMID 24775452
- [Background] Chen KL, Lv ZY, Yang HW, Liu Y, Long FW, Zhou B, Sun XF, Peng ZH, Zhou ZG, Li Y. Effects of Tocilizumab on Experimental Severe Acute Pancreatitis and Associated Acute Lung Injury. Crit Care Med. 2016 Aug;44(8):e664-77. doi: 10.1097/CCM.0000000000001639. PMID 26963319
- [Background] Elcioglu HK, Aslan E, Ahmad S, Alan S, Salva E, Elcioglu OH, Kabasakal L. Tocilizumab's effect on cognitive deficits induced by intracerebroventricular administration of streptozotocin in Alzheimer's model. Mol Cell Biochem. 2016 Sep;420(1-2):21-8. doi: 10.1007/s11010-016-2762-6. Epub 2016 Jul 22. PMID 27443846
- [Background] Araki M, Matsuoka T, Miyamoto K, Kusunoki S, Okamoto T, Murata M, Miyake S, Aranami T, Yamamura T. Efficacy of the anti-IL-6 receptor antibody tocilizumab in neuromyelitis optica: a pilot study. Neurology. 2014 Apr 15;82(15):1302-6. doi: 10.1212/WNL.0000000000000317. Epub 2014 Mar 14. PMID 24634453
- [Background] Ayzenberg I, Kleiter I, Schroder A, Hellwig K, Chan A, Yamamura T, Gold R. Interleukin 6 receptor blockade in patients with neuromyelitis optica nonresponsive to anti-CD20 therapy. JAMA Neurol. 2013 Mar 1;70(3):394-7. doi: 10.1001/jamaneurol.2013.1246. PMID 23358868
- [Background] Ringelstein M, Ayzenberg I, Harmel J, Lauenstein AS, Lensch E, Stogbauer F, Hellwig K, Ellrichmann G, Stettner M, Chan A, Hartung HP, Kieseier B, Gold R, Aktas O, Kleiter I. Long-term Therapy With Interleukin 6 Receptor Blockade in Highly Active Neuromyelitis Optica Spectrum Disorder. JAMA Neurol. 2015 Jul;72(7):756-63. doi: 10.1001/jamaneurol.2015.0533. PMID 25985228
- [Background] Lee WJ, Lee ST, Moon J, Sunwoo JS, Byun JI, Lim JA, Kim TJ, Shin YW, Lee KJ, Jun JS, Lee HS, Kim S, Park KI, Jung KH, Jung KY, Kim M, Lee SK, Chu K. Tocilizumab in Autoimmune Encephalitis Refractory to Rituximab: An Institutional Cohort Study. Neurotherapeutics. 2016 Oct;13(4):824-832. doi: 10.1007/s13311-016-0442-6. PMID 27215218
- [Background] Kleveland O, Kunszt G, Bratlie M, Ueland T, Broch K, Holte E, Michelsen AE, Bendz B, Amundsen BH, Espevik T, Aakhus S, Damas JK, Aukrust P, Wiseth R, Gullestad L. Effect of a single dose of the interleukin-6 receptor antagonist tocilizumab on inflammation and troponin T release in patients with non-ST-elevation myocardial infarction: a double-blind, randomized, placebo-controlled phase 2 trial. Eur Heart J. 2016 Aug 7;37(30):2406-13. doi: 10.1093/eurheartj/ehw171. Epub 2016 May 8. PMID 27161611
- [Derived] Meyer MAS, Bjerre M, Wiberg S, Grand J, Obling LER, Meyer ASP, Josiassen J, Frydland M, Thomsen JH, Frikke-Schmidt R, Kjaergaard J, Hassager C. Modulation of inflammation by treatment with tocilizumab after out-of-hospital cardiac arrest and associations with clinical status, myocardial- and brain injury. Resuscitation. 2023 Mar;184:109676. doi: 10.1016/j.resuscitation.2022.109676. Epub 2022 Dec 24. PMID 36572373
- [Derived] Meyer MAS, Wiberg S, Grand J, Meyer ASP, Obling LER, Frydland M, Thomsen JH, Josiassen J, Moller JE, Kjaergaard J, Hassager C. Treatment Effects of Interleukin-6 Receptor Antibodies for Modulating the Systemic Inflammatory Response After Out-of-Hospital Cardiac Arrest (The IMICA Trial): A Double-Blinded, Placebo-Controlled, Single-Center, Randomized, Clinical Trial. Circulation. 2021 May 11;143(19):1841-1851. doi: 10.1161/CIRCULATIONAHA.120.053318. Epub 2021 Mar 22. PMID 33745292
- [Derived] Meyer MAS, Wiberg S, Grand J, Kjaergaard J, Hassager C. Interleukin-6 Receptor Antibodies for Modulating the Systemic Inflammatory Response after Out-of-Hospital Cardiac Arrest (IMICA): study protocol for a double-blinded, placebo-controlled, single-center, randomized clinical trial. Trials. 2020 Oct 20;21(1):868. doi: 10.1186/s13063-020-04783-4. PMID 33081828